CLINICAL TRIAL: NCT05258838
Title: Tunisian National Registry on Psoriasis
Acronym: PsoTReg
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Société Tunisienne de Dermatologie et de Vénéréologie (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-010-PSOTREG
Record Dates: First submitted 2022-02-14; First posted 2022-02-28 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Psoriasis
Keywords: Psoriasis; Dermatology; Tunisia; Dacima
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
National cross-sectional multicentric study to describe the epidemiological characteristics of patients with Psoriasis in Tunisia

DETAILED DESCRIPTION:
PsoTReg is a Tunisian, descriptive, non-interventional, multicenter and cross-sectional clinical study performed in dermatology departments and outpatients clinics, of both public and private sectors. The study will enroll hospitalized and ambulatory patients with psoriasis disease, by successive inclusions until the end of the recruitment period, set at six months.

A Scientific Committee validates the scientific writing, a Steering Committee supervises the clinical operations of the project.

Collected data are managed by the DACIMA Clinical Suite®, the electronic data capture platform which complies with the FDA 21 CFR part 11 requirements (Food and Drug Administration 21 Code of Federal Regulations part 11), the HIPAA specifications (Health Insurance Portability and Accountability Act), and the ICH standards (International Conference on Harmonisation). A local authorization by the National Agency of Personal Data Protection will be obtained prior to study kick-off.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis
* Informed and written consent

Exclusion Criteria:

* Any dermatology disease other than psoriasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized or outpatient subjects with psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Psoriasis types | At inclusion
  Number of subjects with each type of psoriasis (Plaque psoriasis, Inverse psoriasis, Erythrodermic, Guttate psoriasis, Nail psoriasis, Pustular psoriasis, Psoriatic arthritis)

SECONDARY OUTCOMES:
Demographic | At inclusion
  Demographic data (gender frequency, age mean, body mass index mean) of subjects with psoriasis
Safety assessment of psoriasis medical treatment | At inclusion
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]: Occurrence of infection or tuberculosis or death or any other treatment-related side effect of psoriasis medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Houda Hammami, MD, Study Chair — University Hospital of Habib Thameur, Ben Arous, Tunisia; Mohamed Denguezli, MD, Study Chair — University Hospital of Farhat Hached, Sousse, Tunisia; Asmahen Souissi, MD, Study Director — dr.asmahanesouissi@gmail.com
Locations (1):
- Société Tunisienne de Dermatologie et de Vénéréologie, Tunis, Tunisia, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Facebook page of "Société Tunisienne de Dermatologie et de Vénéréologie" — https://www.facebook.com/stdv.tn/?locale=fr_FR